CLINICAL TRIAL: NCT07200505
Title: A Telerehabilitation Intervention Targeting Core Stability and Muscular Strength in Individuals With Moderate-to-Advanced Hereditary Ataxia: A Pilot Study
Brief Title: Telerehabilitation for Core Stability and Strength in Hereditary Ataxia
Acronym: TRCORE-AH2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat de Lleida (Other)
Responsible Party: Principal Investigator, Maria Masbernat-Almenara, Principal Investigator, Universitat de Lleida
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 25
Record Dates: First submitted 2025-09-12; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Hereditary Ataxia
MeSH Terms: conditions — Spinocerebellar Degenerations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will remain blinded to group allocation. Due to the nature of the intervention, participants and physiotherapists cannot be blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group. TR mixed mode (Experimental): Intervention group: Participants will perform the 12-week exercise program with access to a specially developed telerehabilitation platform. The platform will include videos, questionnaires, a personal diary, automatic reminders, a social chat, and one weekly synchronous supervision session with a physiotherapist to correct technique and adjust progression.
  Interventions: Other: TR Mixed CORE Exercices
- Control group: Asynchronous mode (Active Comparator): Control group: Participants will perform the same exercise program at home but will only receive printed material and videos uploaded to a cloud repository, along with telephone follow-up. They will not have access to the telerehabilitation platform or synchronous sessions.
  Interventions: Other: TR Asyncronous CORE Exercices

INTERVENTIONS:
Other: TR Mixed CORE Exercices — The intervention will last 12 weeks, with five weekly sessions. Prior to starting, all participants will attend three educational sessions and an initial in-person session, during which the physiotherapist will explain and personalise the exercises, ensure proper use of the platform, and provide necessary materials. Participants will then perform the exercises autonomously. he intervention group will receive support through the platform and weekly synchronous supervision, while the control group will only receive basic materials and follow-up phone calls. If needed, family members will be trained to provide occasional assistance with exercise performance.
  Arms: Intervention group. TR mixed mode
Other: TR Asyncronous CORE Exercices — The intervention will last 12 weeks, with five weekly sessions. Prior to starting, all participants will attend three educational sessions and an initial in-person session, during which the physiotherapist will explain and personalize the exercises, ensure proper use of the platform, and provide necessary materials. Participants will then perform the exercises autonomously.
  The intervention group will receive support through the platform and weekly synchronous supervision, while the control group will only receive basic materials and follow-up phone calls. If needed, family members will be trained to provide occasional assistance with exercise performance.
  Arms: Control group: Asynchronous mode

SUMMARY:
This is a two-arm, controlled clinical trial with a parallel design. Participants will be randomly assigned to an intervention or control group. The study is single-blind, as outcome assessors will be blinded to group allocation, while participants and physiotherapists cannot be blinded due to the nature of the intervention. Consecutive sampling will be applied.

For the evaluation of intervention effects (primary and secondary outcomes), the study will follow the Consolidated Standards of Reporting Trials (CONSORT) for non-pharmacological interventions. For the assessment of satisfaction and adherence, a qualitative study will be conducted following the COREQ EQUATOR 17 guidelines to ensure methodological rigor.

The intervention will consist of a 12-week home-based exercise program supervised via mixed telerehabilitation (TR). The control group will perform the same program but receive only telephone follow-up. Four assessments will be conducted: baseline (T0), post-intervention (T1), three months follow-up (T2), and six months follow-up (T3).

DETAILED DESCRIPTION:
This study is a two-arm, controlled, parallel-group clinical trial designed to evaluate the effectiveness, adherence, and satisfaction of a telerehabilitation (TR) program combining core stability and strength exercises with an educational component for people with moderate hereditary ataxia.

Participants will be consecutively recruited through the Catalan Association of Hereditary Ataxias (ACAH), the CSUR Centre for Ataxias and Hereditary Spastic Paraparesis at Hospital Clínic de Barcelona. Eligible participants must have a diagnosis of hereditary spinocerebellar ataxia, moderate severity according to the SARA scale (10-20 points), internet access, basic digital literacy, and provide informed consent.

Participants will be randomly allocated to an intervention or control group. The intervention group will receive three preliminary online educational sessions and then follow a 12-week home-based exercise program delivered through a dedicated telerehabilitation platform. The platform includes pre-recorded videos, weekly synchronous physiotherapy sessions, automated reminders, personal diaries, and interactive features to promote adherence and engagement.

The control group will complete the same 12-week exercise program using printed materials and videos hosted in a cloud repository, supported only by periodic telephone follow-up, without educational sessions or access to the platform.

All participants will undergo four assessments: baseline (T0), post-intervention (T1), and follow-ups at three months (T2) and six months (T3).

The primary outcome is trunk control and sitting balance assessed with the Spanish version of the Trunk Impairment Scale (TIS 2.0). Secondary outcomes include lower limb strength (5x Sit-to-Stand Test), transfer ability (Transfer Assessment Instrument 4.0), upper limb function (Upper Extremity Functional Index), walking speed (4MWT), functional mobility (Timed Up and Go), disease severity (SARA), activities of daily living, health status, falls, adherence (Exercise Adherence Rating Scale and session completion rate), and satisfaction.

Quantitative analyses will follow CONSORT guidelines for non-pharmacological trials, while qualitative data on adherence, satisfaction, perceived risks and benefits, and acceptability will be collected through semi-structured interviews and analyzed thematically according to the COREQ EQUATOR 17 guidelines.

This study will provide evidence on the feasibility, effectiveness, and acceptability of a digital home-based rehabilitation approach for a population with limited access to specialized services, aiming to promote functional autonomy and quality of life while reducing healthcare disparities.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of spinocerebellar hereditary ataxia.
* Moderate severity defined by the SARA scale (10-20 points, Traschütz et al., 2023).
* Stable internet access and suitable electronic devices.

  * Basic digital literacy.
  * Signed informed consent.

Exclusion Criteria:

* Mild (<10) or severe (>20) scores on the SARA scale.
* Severe comorbidities preventing safe exercise participation.
* Severe cognitive impairment that would preclude program adherence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2026-06-12 (Estimated); Study Completion 2026-12-21 (Estimated)

PRIMARY OUTCOMES:
Dynamic sitting balance and coordination | Baseline (T0) , post-intervention (up to 12 weeks), (T1), and follow-ups at 3 months (T2) and 6 months (T3).
  Dynamic sitting balance and coordination will be assessed using the Spanish version of the Trunk Impairment Scale (S-TIS 2.0).
  This scale has a total score range from 0 to 16 points, where higher scores indicate better trunk control, balance, and coordination, and lower scores indicate poorer performance.

SECONDARY OUTCOMES:
Static sitting and standing balance | Baseline (T0), post-intervention (up to 12 weeks)(T1), and follow-ups at 3 months (T2) and 6 months (T3).
  Static sitting and standing balance will be assessed using items 2 and 3 of the Scale for the Assessment and Rating of Ataxia (SARA)
  Item 2 (Stance): scored from 0 to 6 points
  Item 3 (Sitting): scored from 0 to 4 points
  The combined score ranges from 0 to 10 points, where higher scores indicate worse static balance (greater severity of ataxia) and lower scores indicate better balance.
Lower limb functional strength | Baseline (T0) , post-intervention (up to 12 weeks)(T1), and follow-ups at 3 months (T2) and 6 months (T3).
  Assessed using the 5 Times Sit-to-Stand Test (5xSTS). Time in seconds required to stand up and sit down five consecutive times from a standard chair without using the arms.
  Lower scores indicate better performance. Higher scores indicate worse performance.
Transfer ability | Baseline (T0) , post-intervention (up to 12 weeks)(T1), and follow-ups at 3 months (T2) and 6 months (T3).
  Transfer Ability assessed using Transfer Assessment Instrument version 4.0 (TAI 4.0) The TAI 4.0 has a total score range from 0 to 10 points, where higher scores indicate better quality, safety, and independence during transfers and lower scores indicate poorer performance.
Upper limb functionality | Baseline (T0) , post-intervention (up to 12 weeks)(T1), and follow-ups at 3 months (T2) and 6 months (T3).
  Assessed using the Upper Extremity Functional Index (UEFI). The UEFI total score ranges from 0 to 80 points, where higher scores indicate better upper limb function and less difficulty performing daily activities.
Walking Speed | Baseline (T0) , post-intervention (up to 12 weeks)(T1), and follow-ups at 3 months (T2) and 6 months (T3).
  Walking speed, assessed using the 4-Meter Walking Test (4MWT). This test measures the time in seconds needed to walk 4 meters at a comfortable pace. There is no maximum score; shorter times indicate better walking ability, and longer times indicate poorer performance.
Gait Performance | Baseline (T0), post-intervention (up to 12 weeks) (T1), and follow-ups at 3 months (T2) and 6 months (T3)
  Gait performance, assessed using Item 1 (Gait) of the Scale for the Assessment and Rating of Ataxia (SARA).
  This item is scored from 0 to 8 points, where higher scores indicate worse gait performance (greater severity of ataxia) and lower scores indicate better gait.
Functional mobility and fall risk | Baseline (T0) , post-intervention (up to 12 weeks)(T1), and follow-ups at 3 months (T2) and 6 months (T3).
  Assessed using the Timed Up and Go Test (TUG). This test measures the time in seconds needed to stand up from a chair, walk 3 meters, turn around, return, and sit down.
  There is no maximum score; shorter times indicate better mobility and lower fall risk, and longer times indicate worse mobility and higher fall risk.
Disease severity | Baseline (T0) , post-intervention (up to 12 weeks)(T1), and follow-ups at 3 months (T2) and 6 months (T3).
  Assessed using Scale for the Assessment and Rating of Ataxia (SARA). The SARA has a total score range from 0 to 40 points, where higher scores indicate greater severity of ataxia and lower scores indicate less severe symptoms.
Program Compliance | Post-intervention (up to 12 weeks)(T1), and follow-ups at 3 months (T2) and 6 months (T3).
  Program compliance will be assessed using the percentage of completed prescribed sessions, calculated as: (number of minutes or exercises completed / number prescribed) × 100. Higher percentages indicate greater compliance, while lower percentages indicate poorer compliance.
Exercise Adherence | Post-intervention (up to 12 weeks) (T1), and follow-ups at 3 months (T2) and 6 months (T3).
  Exercise adherence assessed using Exercise Adherence Rating Scale (EARS) The EARS has a total score range from 0 to 24 points, where higher scores indicate better adherence to the exercise program.
Satisfaction, perceived benefits, risks, and acceptability | Post-intervention (up to 12 weeks)(T1)
  Participant satisfaction, perceived benefits, risks, barriers, and overall acceptability of the program will be assessed through semi-structured interviews conducted after completing the intervention. Interviews will last approximately 45 minutes and will be analyzed using thematic content analysis following COREQ guidelines.
  This is a qualitative outcome without a numerical score.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Masbernat-Almenara, Principal Investigator — Universitat de Lleida; Selma Pelàez Hervàs, Study Chair — Hospital Clinic of Barcelona; Helena Fernández Lago, Study Chair — Universitat de Lleida
Locations (1):
- University of Lleida, Lleida, Lleida, Spain

IPD SHARING:
Plan to Share IPD: Yes
IPD will be made available in open access at the Catalan Open Research Area (CORA) repository, in accordance with the FAIR data principles and current data protection regulations (EU GDPR and Spanish Organic Law 3/2018). De-identified datasets will be deposited after publication of the main study results and will be accessible to other researchers upon reasonable request through the CORA platform.
Time Frame: Data will be available within 12 months after publication of the main study results and will remain accessible for at least 5 years.
Access Criteria: Access will be granted to researchers upon reasonable request through the CORA platform. Requests must include a short proposal describing the intended use of the data and will be reviewed by the study's principal investigator and steering committee. Data will only be used for scientific purposes aligned with the consent provided by participants.
  Data sheets will be openly accessible through the CORA platform without restriction.
URL: https://dataverse.csuc.cat/